CLINICAL TRIAL: NCT00750789
Title: The Effect of Dates on Plasma Lipids, Oxidative Stress and the Atherogenicity of Serum in Healthy Adults
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Wasseem Rock, emek medical center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 0061-08-EMC
Record Dates: First submitted 2008-08-17; First posted 2008-09-11 (Estimated); Last update posted 2008-09-11 (Estimated); Status verified 2008-09

CONDITIONS: Atherosclerosis
MeSH Terms: conditions — Atherosclerosis | interventions — Chronology as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Dietary Supplement: dates — 5 maedjool dates or 7 emery dates per day for 2 weeks each with a washout period of 2 weeks between

SUMMARY:
It has been proven in in-vitro studies that dates decrease the oxidative stress in serum. There have been no in-vivo studies to this date. The current study aims to test whether dates consumption by healthy adults decreases serum oxidative stress and improves serum PON1 activity and serum lipid profile.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2008-09; Primary Completion 2008-11 (Estimated)

PRIMARY OUTCOMES:
serum oxidative stress | 30 days

SECONDARY OUTCOMES:
serum lipid profile | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Wasseem Rock, Principal Investigator — Emek Medical Center
Locations (1):
- Emek Medical Center, Afula, Israel